CLINICAL TRIAL: NCT02555306
Title: A Phase I/II, Open-label, Dose-escalating, Sequential-cohort Study Assessing the Safety, Tolerability, Immunogenicity, and Bioactivity of a Single Intravitreal Injection of DE-122 Injectable Solution for the Treatment of Refractory Exudative Age-related Macular Degeneration
Brief Title: A Phase I/II Safety, Tolerability, Immunogenicity, and Bioactivity Study of DE-122 Injectable Solution for Refractory Exudative Age-related Macular Degeneration
Acronym: PAVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36-001
Record Dates: First submitted 2015-09-13; First posted 2015-09-21 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Dose DE-122 (Experimental): Single intravitreal injection of DE-122 Low Dose Injectable Solution
  Interventions: Drug: 0.5 mg of DE-122
- Medium-Low Dose DE-122 (Experimental): Single intravitreal injection of DE-122 Medium-Low Dose Injectable Solution
  Interventions: Drug: 1.0 mg of DE-122
- Medium-High Dose DE-122 (Experimental): Single intravitreal injection of DE-122 Medium-High Dose Injectable Solution
  Interventions: Drug: 2.0 mg of DE-122
- High Dose DE-122 (Experimental): Single intravitreal injection of DE-122 High Dose Injectable Solution
  Interventions: Drug: 4.0 mg of DE-122

INTERVENTIONS:
Drug: 0.5 mg of DE-122 — DE-122 Injectable Solution
  Arms: Low Dose DE-122
Drug: 1.0 mg of DE-122 — DE-122 Injectable Solution
  Arms: Medium-Low Dose DE-122
Drug: 2.0 mg of DE-122 — DE-122 Injectable Solution
  Arms: Medium-High Dose DE-122
Drug: 4.0 mg of DE-122 — DE-122 Injectable Solution
  Arms: High Dose DE-122

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, immunogenicity, and bioactivity of a single intravitreal (IVT) administration of DE-122 in subjects with refractory exudative age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent
* Diagnosis of subretinal or intraretinal fluid secondary to exudative age-related macular degeneration
* Prior treatment in the study eye with any intravitreal anti-VEGF medication
* At least one lesion in the study eye that meets minimal pathology criteria
* Best corrected visual acuity of 65 to 20 ETDRS letters in the study eye
* Best corrected visual acuity of 20/200 or better in the fellow eye
* Reasonably clear media and some fixation in the study eye

Exclusion Criteria:

Ocular

* Use or anticipated use of any intravitreal, periocular or photodynamic therapy in the study eye for the treatment of AMD within a specified timeframe prior to Visit 1
* Uncontrolled or advanced glaucoma, chronic hypotony or vitrectomy in the study eye
* Evidence of any other ocular disease other than exudative age-related macular degeneration in the study eye that may confound the outcome of the study
* Need for ocular surgery in the study eye during the course of the study
* Presence or history of certain ocular or periocular pathology or conditions that could limit the ability to perform required study assessments in either eye and/or confound study results

Non-Ocular

* Allergy or hypersensitivity to study drug product, fluorescein dye or other study-related procedures and medications
* Current or history of certain systemic conditions, abnormalities or therapies that would render a subject a poor candidate for the study
* Participation in other investigational drug or device clinical trials within 30 days prior to randomization or planning to participate in other investigational drug or device clinical trials for the duration of the study
* Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions and men who do not agree to practice an acceptable method of contraception throughout the course of the study
* Unable to comply with study procedures or follow-up visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mountain View, California
  - Walnut Creek, California
  - Jackson, Michigan
  - Austin, Texas
  - McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5 mg of DE-122: Single intravitreal injection of Low Dose DE-122 Injectable Solution
- 1.0 mg of DE-122: Single intravitreal injection of Medium-Low Dose DE-122 Injectable Solution
- 2.0 mg of DE-122: Single intravitreal injection of Medium-High Dose DE-122 Injectable Solution
- 4.0 mg of DE-122: Single intravitreal injection of High Dose DE-122 Injectable Solution
Period: Overall Study
Arm/Group | 0.5 mg of DE-122 | 1.0 mg of DE-122 | 2.0 mg of DE-122 | 4.0 mg of DE-122
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg of DE-122 | 1.0 mg of DE-122 | 2.0 mg of DE-122 | 4.0 mg of DE-122 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 2 | 3 | 3 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (4.2) | 73.7 (1.2) | 74.0 (6.2) | 84.0 (7.2) | 74.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 2 | 7
  Male | 0 | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Day 90.
Description: BCVA measures the acuteness or clearness of best-corrected vision in ETDRS (Early Treatment of Diabetic Retinopathy Study) letters, with a range of [0, 97] in ETDRS letters.
  An increase in BCVA indicates an improvement in the best corrected vision.
Time Frame: Baseline (Day1) and Day 90.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | 0.5 mg of DE-122 | 1.0 mg of DE-122 | 2.0 mg of DE-122 | 4.0 mg of DE-122
Number analyzed (Participants) | 3 | 3 | 3 | 3
ETDRS letters | -1.3 (2.1) | 2.7 (5.0) | 1.0 (7.9) | 3.3 (4.5)

2. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST) at Day 90.
Description: Bioactivity measures include CST (μm) measured by SD-OCT. Bioactivity will be considered evident if a considerable decrease in CST is observed.
Time Frame: Baseline (Day1) and Day 90.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | 0.5 mg of DE-122 | 1.0 mg of DE-122 | 2.0 mg of DE-122 | 4.0 mg of DE-122
Number analyzed (Participants) | 3 | 3 | 3 | 3
microns | -116.3 (194.9) | 62.7 (68.1) | -36.0 (42.6) | -111.3 (171.2)

ADVERSE EVENTS:
Time Frame: From Visit 1 (Day 1) to Study Exit (Day 90)]
Groups:
- 0.5 mg of DE-122: Single intravitreal injection of Low Dose DE-122
- 1.0 mg of DE-122: Single intravitreal injection of Medium-Low Dose DE-122
- 2.0 mg of DE-122: Single intravitreal injection of Medium-High Dose DE-122
- 4.0 mg of DE-122: Single intravitreal injection of High Dose DE-122
Arm/Group | 0.5 mg of DE-122 | 1.0 mg of DE-122 | 2.0 mg of DE-122 | 4.0 mg of DE-122
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg of DE-122 (N=3) | 1.0 mg of DE-122 (N=3) | 2.0 mg of DE-122 (N=3) | 4.0 mg of DE-122 (N=3)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Deposit eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyphaema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02555306/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02555306/SAP_001.pdf